CLINICAL TRIAL: NCT05265715
Title: A Low AGE (Advanced Glycation End-product) Dietary Intervention for Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202201100
Record Dates: First submitted 2022-01-31; First posted 2022-03-03 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low AGE dietary intervention (Experimental): * Patients will complete a food frequency questionnaire, & if found to have a high AGE diet at baseline, will then begin the study the 24-week low AGE dietary intervention. Patients will complete a 3 day food record prior to receiving remotely delivered education on AGEs on how to adhere to a low AGE diet by the study dieticians prior to starting. This session will provide education on dietary AGE & how to prepare & choose low AGE meals
  * Subsequent sessions with the dieticians will be conducted remotely & will be 30-60 minutes in duration, with the exception of sessions scheduled for weeks when a study blood draw is required, when visits with the dietician may occur in person. These sessions will occur at the following schedule: weekly during the first 2 months (8 sessions), every other week during the next 2 months (4 sessions, aka step down sessions), monthly for the remaining 2 months (2 sessions)
  * 3 day food records will be collected at 12 & 24 weeks, in addition to baseline.
  Interventions: Other: Low AGE diet; Procedure: Research blood draw

INTERVENTIONS:
Other: Low AGE diet — The recommended daily AGE intake will be either:
  * 7,500 kilounits [ku], which is a 50% reduction from the average 15,000 ku consumed by most adults or
  * a 50% reduction from their baseline AGE intake (based on 3-day food AGE record)
Procedure: Research blood draw — Baseline (Week 0), Week 4, Week 12, and Week 24 (end of intervention)

SUMMARY:
The scientific premise for this study is the known impact of overweight/obesity on breast cancer risk and outcomes, the association between advanced glycation end-products (AGE) and high fat, highly processed foods common in Western diets, and the preclinical evidence suggesting a link between AGE and breast cancer independent of weight. The association between dietary and serum AGE in breast cancer survivors and prognosis has not been previously evaluated. However, preclinical studies suggest that AGE may represent a novel, lifestyle-linked, modifiable, prognostic biomarker, which could be targeted through lifestyle (diet and exercise) and/or pharmaceutical interventions to improve breast cancer prognosis. The proposed study will pave the way for a large scale randomized controlled trial to evaluate the impact of a low AGE diet on weight (BMI), known (IL-6 and CRP) and novel (AGE and RAGE) prognostic biomarkers, and ultimately on breast cancer prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer, any subtype, stage I-III, within the last 36 months, who have completed primary therapy of their breast cancer (surgery, radiation, and chemotherapy). Must be at least 4 weeks post their last chemotherapy or radiation therapy. Concurrent hormonal therapy is allowed.
* At least 18 years of age.
* Determined to have a high AGE diet at baseline (dietary AGE intake greater than 14 Eq/day as assessed by food frequency questionnaire).
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Diagnosis of diabetes.
* History of eating disorder or body dysmorphic disorder.
* Active tobacco use (tobacco is a source of advanced glycation end products).
* Active participation in other dietary or physical activity clinical trials or community interventions.
* Taking and unwilling/unable to stop taking B-6 (pyridoxamine), B1 (thiamine) or metformin (all known AGE inhibitors).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by adherence rate | At study completion for all enrolled participants (estimated to be 15 months)
  * Feasibility is a defined adherence rate of at least 80% of participants enrolled
  * Diet adherence will be categorized by the study dietitian at the end of the study and before the results of AGEs in serum or any analysis of outcomes to avoid bias. Following each phone session with the participants, the dietitian will elicit answers to the following question: since the last call did the participant use any cooking methods they were advised to avoid for certain food items? (yes/no).
  * The information will be used to calculate an adherence score. Adherence score is % phone calls of patient's report for full maintaining instructions to reduce AGEs.
  * Very high adherence= ≥80%; good adherence= 60-80%; partial adherence= 40-60%; lack of adherence but intention to adhere more in the future= ≤40%; lack of adherence and no intention to adhere more= ≤40%
Feasibility as measured by dropout rate | At study completion for all enrolled participants (estimated to be 15 months)
  -Feasibility is defined as a dropout rate of less than 20% of participants enrolled

SECONDARY OUTCOMES:
Change in dietary AGE | At baseline and study completion (24 weeks)
  -Dietary AGE is estimated based on analysis of the 3 day food record patients will complete at baseline and study completion. A specific dietary AGE value will be assigned to each item on the 3 day food recall by consultant and dietary AGE expert Jaime Uribarri, MD. This value is based on his published dietary AGE database which accounts for type of food, portion size and cooking methods.
Change in serum AGE | Baseline, week 12, and week 24
  * Blood specimens for serum AGE analysis will be shipped from the University of San Diego Biorepository to the Medical University of South Carolina to be analyzed in the lab of study team member and expert AGE analyst, Dr. David Turner.
  * AGE (measured by the AGE metabolite carboxymethyllysine (ug/ml)) will be assessed in serum using commercially available 96-well format ELISA's and ROS detection kits (Cell Biolabs). Nε-carboxymethyllysine (CML) is an AGE metabolite extensively studied in animal models of disease and with regard to food content.
Correlation between serum AGE levels and BMI | Baseline, 12 weeks, and 24 weeks
  -The relationship between serum AGE levels and BMI will be assessed using rank based correlation.
Correlation between serum AGE levels and serum CRP | Baseline, 12 weeks, and 24 weeks
  -The relationship between serum AGE levels and serum CRP will be assessed using rank based correlation.
Correlation between serum AGE levels and IL6 | Baseline, 12 weeks, and 24 weeks
  -The relationship between serum AGE levels and IL6 will be assessed using rank based correlation.
Correlation between serum AGE levels and glucose | Baseline, 12 weeks, and 24 weeks
  -The relationship between serum AGE levels and glucose will be assessed using rank based correlation.
Correlation between serum AGE levels and leptin | Baseline, 12 weeks, and 24 weeks
  -The relationship between serum AGE levels and leptin will be assessed using rank based correlation.
Correlation between serum AGE levels and adiponectin | Baseline, 12 weeks, and 24 weeks
  -The relationship between serum AGE levels and adiponectin will be assessed using rank based correlation.
Correlation between dietary AGE and BMI | Baseline, 12 weeks, and 24 weeks
  -The relationship between dietary AGE and BMI will be assessed using rank based correlation.
Correlation between dietary AGE and serum CRP | Baseline, 12 weeks, and 24 weeks
  -The relationship between dietary AGE and serum CRP will be assessed using rank based correlation.
Correlation between dietary AGE and IL6 | Baseline, 12 weeks, and 24 weeks
  -The relationship between dietary AGE and IL6 will be assessed using rank based correlation.
Correlation between dietary AGE and insulin | Baseline, 12 weeks, and 24 weeks
  -The relationship between dietary AGE and insulin will be assessed using rank based correlation.
Correlation between dietary AGE and glucose | Baseline, 12 weeks, and 24 weeks
  -The relationship between dietary AGE and glucose will be assessed using rank based correlation.
Correlation between dietary AGE and leptin | Baseline, 12 weeks, and 24 weeks
  -The relationship between dietary AGE and leptin will be assessed using rank based correlation.
Correlation between dietary AGE and adiponectin | Baseline, 12 weeks, and 24 weeks
  -The relationship between dietary AGE and adiponectin will be assessed using rank based correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Peterson, M.D., MSCR, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
All research data will be shared between Dr. Peterson and the study team will be available to all investigators named on this proposal. The primary investigators are also willing to share data and materials with other eligible investigators and collaborators through academically established means. Final data will be shared in an openly and timely manner while ensuring the privacy and confidentiality of participants through presentations at scientific seminars and conference and publications in peer reviewed journals. Information about the intervention protocol and survey tools will be made available to others upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article presentation.
Access Criteria: Proposals should be directed to llpeterson@wustl.edu.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu